CLINICAL TRIAL: NCT03514381
Title: Pharmacologic Interaction Between Ifosfamide and Aprepitant in Treated Patients With Soft Tissue Sarcoma
Acronym: IPIAP-STM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17 SARC 04
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; Ifosfamide; Aprepitant; Doxorubicin
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients starting a treatment with Doxorubicin and Ifosfamide (Other)
  Interventions: Drug: Patients starting a treatment with Doxorubicin and Ifosfamide

INTERVENTIONS:
Drug: Patients starting a treatment with Doxorubicin and Ifosfamide — 9 blood samples will be collected at each Cycle:
  * Cycle 1 (Day 1-Day 2-Day 3)
  * Cycle 2 (Day 1-Day 2-Day 3)

SUMMARY:
This trial is a multicentric study aiming to assess the evolution of the serum ifosfamide concentrations and its serum metabolites in patients treated for an Soft Tissue Sarcoma and co-exposed to Aprepitant.

The study will be conducted on a population of patients treated with Doxorubicin and Ifosfamide. The Aprepitant can be prescribed to patients from cycle 2, according to the current recommendations. Doxorubicin, Ifosfamide and Aprepitant will be administered in the context of routine care. The follow-up during the treatment period and the clinical, biological and radiological assessments will be performed according to the standard of each centre.

Patients will be followed during the two first cycles of treatment. For the pharmacokinetic study, blood samples will be collected at different time points during the 2 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Anatomopathologic diagnosis of soft tissue sarcoma (localized, local recidive or metastatic).
3. Patient receiving doxorubicin and ifosfamide chemotherapy (treatment decided during Multidisciplinary consultation meetings) (neoadjuvant, adjuvant or palliative treatment).
4. Screening laboratory values must meet the following criteria:

   1. Hemoglobin > 9.0 g/dL, Neutrophils > 1500/mm3, Platelets > 100000/mm3
   2. Creatinine clearance (MDRD formula) > 60ml/min.
   3. AST/ALT < 2.5 x ULN (5 x ULN in patients with hepatic metastasis).
5. Evaluable disease (measurable per RECIST or not), if applicable.
6. Patient must provide written informed consent prior to any study specific procedures.
7. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Previous treatment with Ifosfamide.
2. Patient who has already started doxorubicin and ifosfamide treatment.
3. Any medical condition that can increase the patient's risk

   1. Active infection
   2. Active hepatitis or cirrhosis
   3. Recipients of organ transplants or immunocompromised patients, including Human Immunodeficiency Virus (HIV) infection
4. Pregnant or breastfeeding women
5. Any psychological, familial, geographical or sociological condition which does not allow to respect the medical follow-up and/or compliance to study procedure
6. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Evolution of 2d-Ifo plasma concentrations between the 1st cycle (without co-exposure to the Aprepitant) and the 2nd cycle (with co-exposure to the Aprepitant) | Cycle 2 Day 3 for each patient

SECONDARY OUTCOMES:
Toxicity assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 | Cycle 3 Day 1 for each patient
Evolution of plasma concentrations of ifosfamide and its serum metabolites between the first and second cycles | Cycle 3 Day 1 for each patient
The rate of objective responses determined according to the criteria RECIST v 1.1 | Cycle 3 Day 1 for each patient

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut Bergonie, Bordeaux
  - Institut Regional Du Cancer de Montpellier (Icm), Montpellier
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse